CLINICAL TRIAL: NCT06574412
Title: The Efficacy and Safety of Cardonilizumab Combined With Lenvastinib in Perioperative Treatment of Resectable Renal Clear Cell Carcinoma-A Single-arm, Single-center, Exploratory Clinical Study
Brief Title: Cardenilimab Combined With Lenvatinib in Patients With Perioperative Resectable Clear Cell Renal Cell Carcinoma.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ziling Liu, Principal Investigator, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-HS-091
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Resectable Clear Cell Carcinoma of the Kidney

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant -surgery-adjuvant therapy group (Experimental): Preoperative: Cardenilimab was administered at a dose of 10 mg/kg intravenously once daily, with one cycle every 21 days, for a total of 4 cycles. Lenvatinib was prescribed as follows: for patients weighing less than 60 kg, 8 mg was given orally once daily for 4 cycles; for those weighing more than 60 kg, 12 mg was administered orally once daily for a total of 4 cycles. Surgery: The patient underwent standard radical nephrectomy 30 to 40 days after completing the 4 cycles of lenvatinib treatment. Postoperative: Cardenilimab was continued at a dose of 10 mg/kg intravenously once daily, with one cycle every 21 days, for a total of 8 cycles. Lenvatinib dosing postoperatively was as follows: for patients weighing less than 60 kg, 8 mg was given orally once daily for a total of 8 cycles; for those weighing more than 60 kg, 12 mg was administered orally once daily for a total of 8 cycles.
  Interventions: Drug: cardonilizumab combined with renvastinib

INTERVENTIONS:
Drug: cardonilizumab combined with renvastinib — Preoperative: Cardenilimab: 10 mg/kg qd intravenously, one cycle every 21 days, administered on the first day of each cycle, a total of 4 cycles. Lenvatinib: Weight <60kg, 8mg, once a day, orally, for 4 cycles Weight >60kg, 12mg, once a day, orally, for a total of 4 cycles Surgery: The patient is receiving 4 cycles of cardenilimab + Standard radical nephrectomy was performed within 30-40 days after the end of lenvatinib treatment. Postoperative: Cardenilimab: 10 mg/kg qd intravenously, 1 cycle every 21 days, administered on the 1st day of each cycle, a total of 8 cycles Lenvatinib: body weight <60 kg, 8 mg, once a day, orally , a total of 8 cycles, weight > 60kg, 12mg, once a day, orally, a total of 8 cycles.

SUMMARY:
This study is a single-arm, single-center, phase II clinical study. The main purpose is to evaluate the perioperative efficacy and safety of cardenilimab combined with lenvatinib in patients with resectable clear cell renal cell carcinoma. This study included a screening period, a treatment period, and a follow-up period. After completing the examination and assessment during the screening period, qualified subjects will enter the study treatment period after signing the informed consent form. Subjects should receive induction therapy and maintenance therapy in accordance with the protocol until there is disease progression on imaging as judged by the investigator based on RECIST 1.1 standards, intolerable toxicity, or the subject voluntarily requests to terminate study treatment or withdraws information. Agree, or the researcher determines that treatment needs to be terminated. (1) Primary research endpoint: Objective response rate (ORR) of primary tumor according to RECIST 1.1 criteria (2) Secondary research endpoint: 1. According to RECIST 1.1, as assessed by the investigator: (1) Progression-free survival (Progress Free Survival, PFS); (2) Overall survival (OS); 2. Type, incidence and severity of adverse events (AE) and serious adverse events (SAE) assessed in accordance with NCI-CTCAE 5.0 . 3. Pathological response rate (MPR), R0 resection rate 4. Based on Quality of Life QoL score.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients: 18-75 years old;
2. ECOG physical condition score: 0~2 points;
3. Histologically confirmed resectable non-metastatic clear cell carcinoma of the kidney (TNM staging criteria for renal carcinoma);
4. Expected survival ≥12 weeks;
5. Have not received systemic anti-tumor therapy before;
6. Major organ function is normal, that is, relevant examination indicators within 14 days before randomization meet the following requirements: 1) Blood routine examination: a) hemoglobin ≥90 g/L (no blood transfusion within 14 days); b) Neutrophil count ≥1.5×109/L; c) Platelet count ≥100×109/L; 2) Biochemical examination: a) Total bilirubin ≤ 1.5×ULN (upper limit of normal value); b) Serum glutamic-pyruvic aminotransferase (ALT) or serum glutamic-oxalic aminotransferase (AST) ≤ 2.5×ULN; If there is liver metastasis, ALT or AST ≤ 5×ULN; c) Serum creatinine <1.5 times the upper limit of normal; Endogenous creatinine clearance ≥ 50 ml/min (Cockcroft-Gault formula); 3) Routine coagulation test: a) International Standardized ratio (INR) or prothrombin time (PT) ≤1.5 X ULN. b) Activated partial thromboplastin time (APTT) ≤1.5 x ULN. 4) Cardiac Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ 50%.
7. Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days prior to inclusion, with a negative result, and be willing to use an appropriate method of contraception during the test period and for 8 weeks after the last dose of the test drug. For men, consent to use appropriate methods of contraception or surgical sterilization during the trial period and within 8 weeks after the last dose of the trial drug;
8. The subjects voluntarily joined the study and signed the informed consent, with good compliance and follow-up.

Exclusion Criteria:

1. Other malignancies diagnosed within 5 years prior to administration, excluding radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ. If another malignant tumor or lung cancer is diagnosed more than 5 years before administration, pathological or cytological diagnosis of recurrent lesions is required.
2. Currently participating in an interventional clinical study or receiving other drugs or investigational devices within 4 weeks prior to initial dosing;
3. Previous treatment with anti-PD-1, anti-PD-L1 or anti-PD-L2 drugs or drugs that target another stimulus or synergistically inhibit T cell receptors (e.g. CTLA-4, OX-40, CD137);
4. Received immunomodulatory drugs (thymosin, interferon, interleukin, etc.) within 2 weeks before the first dose, or received major surgical treatment within 3 weeks before the first dose;
5. Have a history of bleeding, any bleeding event with a severity rating of CTCAE5.0 or higher occurring within 4 weeks prior to screening;
6. Received solid organ or blood system transplantation;
7. Clinically uncontrolled active infections, including but not limited to acute pneumonia;
8. History of idiopathic pulmonary fibrosis, institutional pneumonia (such as bronchiolitis obliterans), and drug-related pneumonia;
9. Uncontrolled or symptomatic hypercalcemia; 10.III-IV and congestive heart failure (New York Heart Association classification), poorly controlled and clinically significant arrhythmias;
10. Known allergic reactions to PD-1 monoclonal antibody, albumin paclitaxel, carboplatin active ingredients and/or any excipients;
11. An active autoimmune disease requiring systemic treatment (e.g. with disease-modifying drugs, corticosteroids, or immunosuppressants) has occurred within 2 years prior to first administration. Replacement therapies (such as thyroxine, insulin, or physiological doses of corticosteroids for adrenal or pituitary insufficiency) are not considered systemic；
12. Patients requiring long-term systemic use of corticosteroids. Patients with COPD or asthma requiring intermittent use of bronchodilators, inhaled corticosteroids, or local injections of corticosteroids could be enrolled；
13. Wounds that have not healed for a long time or fractures that have not healed completely;
14. Have an active infection requiring treatment or have used systemic anti-infective drugs within 1 week prior to first dosing;
15. Arterial thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), myocardial infarction, and unstable angina pectoris, occurred within 6 months before screening;
16. Known history of human immunodeficiency virus (HIV) infection (i.e., HIV1/2 antibody positive);
17. Untreated active hepatitis B; Note: Hepatitis B subjects who meet the following criteria are also eligible for inclusion: HBV viral load must be < 1000 copies /ml (200IU/ml) prior to initial dosing, and subjects should receive anti-HBV therapy to avoid viral reactivation throughout the duration of study chemotherapy drug treatment. For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required.
18. Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower limit of detection)
19. Those who have a history of psychotropic drug abuse and cannot quit or have mental disorders;
20. Have received live vaccine within 30 days prior to the first dose;Note: Injectable inactivated virus vaccine against seasonal influenza is permitted; However, live attenuated influenza vaccines administered intranasally are not permitted.
21. There is a medical history, illness, treatment, or abnormal laboratory result that could interfere with the test results or prevent the subject from fully participating in the study, or the investigator believes that participation in the study is not in the subject's best interest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
ObjectiveResponse Rate，ORR | The proportion of patients whose tumor size reduction reaches predetermined limits and persists over
  Objective Response Rate was defined as the percentage of participants with a complete response (CR) or partial response (PR)

SECONDARY OUTCOMES:
Overall survival，OS | The time from randomization to death (from any cause)
  OS was defined as the time from the first study treatment to the date of death from any cause
Progress Free Survival，PFS | The time between the start of randomization and the progression of tumor development (in any respect
  PFS was defined as the time from randomization to tumor progression (any aspect) or death (from any cause).
Types, incidence, and severity of adverse event (AE) | 28 days after the last dose of study treatment
  Classification per Common Terminology Criteria for Adverse Events (CTC-AE) version 5.0.
Types, incidence, and severity of serious adverse event (SAE) | 28 days after the last dose of study treatment
  Classification per Common Terminology Criteria for Adverse Events (CTC-AE) version 5.0.
major pathologic response, MPR | After neoadjuvant therapy, the percentage of surviving tumor cells in the tumor bed was less than 10
After neoadjuvant therapy, the percentage of surviving tumor cells in the tumor bed was less than 10 | Standard radical nephrectomy
Quality of life score | 28 days after the last dose of study treatment
  Classified according to EORTC QLQ-C30 (V3.0 Chinese Version).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] [1] Siegel RL, Miller KD, Jemal A: Cancer statistics, 20182018;68: 7-30. [2] 赫捷．2018 中国肿瘤登记年报［Ｍ］．北京：人民卫生出 版社，2019：129 [3] Motzer RJ, Hutson TE, Tomczak P, et al. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma [J]. N Engl J Med, 2007, 356(2): 115-124. [4] Escudier B, Szczylik C, Hutson T E, et al. Randomized phase II trial of first-line treatment with sorafenib versus interferon Alfa-2a in patients with metastatic renal cell carcinoma [J]. Journal of clinical oncology, 2009, 27(8): 1280-1289. [5] Motzer R J, Hutson T E, Tomczak P, et al. Sunitinib versus interferon alfa in metastatic renal-cell carcinoma [J]. New England Journal of Medicine, 2007, 356(2): 115-24. [6] 韩雪冰.靶向联合免疫治疗提高晚期肾癌疗效[J].健康向导,2023,29(01):15. [7] 张凯,朱刚．2020 版 EAU 肾细胞癌诊疗指南更新解读 之二［J］．中华泌尿外科杂 2020， 41( 8) : 578-580． [8] 邓 建 华 , 纪 志 刚 . 高 危 肾 细 胞 癌 术 前 新 辅 助 靶 向 药 物 治 疗 [J]. 现 代 泌 尿 外 科 杂 志,2018,23(06):405-408. [9] 李凡,管维.肾癌诊疗相关进展[J].临床外科杂志,2021,29(02):101-104. [10] Bex A, van Thienen JV, Schrier M, et al. A Phase II, single-arm trial of neoadjuvant axitinib plus avelumab in patients with localized renal cell carcinoma who are at high risk of relapse after nephrectomy (NEOAVAX) [published correction appears in Future Oncol. 2019 Aug;15(22):2667]. Future Oncol. 2019;15(19):2203-2209. [11] Karam JA, Msaouel P, Haymaker CL, Matin SF, Campbell MT, Zurita AJ, Shah AY, Wistuba II, Marmonti E, Duose DY, Parra ER, Soto LMS, Laberiano-Fernandez C, Lozano M, Abraham A, Hallin M, Chin CD, Olson P, Der-Torossian H, Yan X, Tannir NM, Wood CG. Phase II trial of neoadjuvant sitravatinib plus nivolumab in patients undergoing nephrectomy for locally advanced clear cell renal cell carcinoma. Nat Commun. 2023 May 10;14(1):2684.